CLINICAL TRIAL: NCT01627301
Title: Mechanisms of Sympathetic Overactivity in Post-traumatic Stress Disorder
Brief Title: Sympathetic Overactivity in Post-traumatic Stress Disorder
Acronym: SO-PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jeanie Park, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00054697; 2025P011325 (Other: Emory IRB)
Record Dates: First submitted 2012-06-21; First posted 2012-06-25 (Estimated); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Post-traumatic Stress Disorder; Prehypertension
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Prehypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Device-guided Breathing (DGB) (Experimental): Participants randomized to the DGB group use a device to guide their breathing to a slow breathing rate.
  Interventions: Device: Device-Guided Breathing (DGB)
- Sham DGB (Sham Comparator): Participants randomized to the sham DGB group use a device identical to the DGB device but respiratory rates are not guided lower than the physiological rate.
  Interventions: Device: Sham DGB
- Transcutaneous Vagal Nerve Stimulation (tVNS) (Experimental): Participants randomized to use a tVNS device to deliver mild electrical stimulation to the vagal nerve.
  Interventions: Device: Transcutaneous Vagal Nerve Stimulation (tVNS)
- Sham tVNS (Sham Comparator): Participants randomized to use the sham tVNS device which vibrates but does not stimulate the vagal nerve.
  Interventions: Device: Sham tVNS

INTERVENTIONS:
Device: Device-Guided Breathing (DGB) — The RESPeRATE device will be used for 15 minutes of device-guided breathing daily for 8 weeks. The participant places the elastic belt with a respiration sensor around the upper abdomen, and wears earbuds for audio feedback. The device monitors the breathing rate, calculates inspiration and expiration times, and generates a personalized melody of two distinct ascending and descending tones for inhalation versus exhalation. Users effortlessly entrain their breathing pattern with the tones, and the device gradually guides the user to a prolonged expiration time and slower respiratory rate (to < 10 breaths/minute). The device automatically stores usage data, allowing for quantification of adherence and performance.
  Other Names: RESPeRATE
  Arms: Device-guided Breathing (DGB)
Device: Sham DGB — The sham device is identical to the DGB device, except it does not guide respiratory rates to slow down and instead maintains a rate of 14 breaths per minute. The sham device is used for 15 minutes per day for 8 weeks.
  Arms: Sham DGB
Device: Transcutaneous Vagal Nerve Stimulation (tVNS) — tVNS is a noninvasive method that involves placing a device over the skin overlying the vagus nerve on the neck. The device delivers mild electrical stimulation, using transcutaneous electrical nerve stimulation (TENS) unit. The stimulation is increased until there is a vibration and slight muscle contraction in the lower face or neck. Then the stimulation is delivered for 2 minutes on the left side of the neck, and on the right side of the neck, for a total of 4 minutes. The tVNS device is used twice daily for 8 weeks.
  Other Names: gammaCore
  Arms: Transcutaneous Vagal Nerve Stimulation (tVNS)
Device: Sham tVNS — Sham stimulation is delivered using a device that is identical to the gammaCore device but is programed to deliver a lower frequency that can be felt by the participant but does not actually stimulate the vagus nerve. The sham device is used twice daily for 8 weeks.
  Arms: Sham tVNS

SUMMARY:
Post-traumatic stress disorder (PTSD) is a highly prevalent anxiety disorder that is associated with an increased risk of cardiovascular (CV) disease and hypertension. One potential mechanism is overactivation of the sympathetic nervous system (SNS), both at rest and particularly during stress. This study will evaluate whether 8 weeks of daily DGB therapy or transcutaneous vagus nerve stimulation (tVNS) therapy improves SNS activity at rest and during stress.

DETAILED DESCRIPTION:
PTSD is highly prevalent in both the military and general population. Because of the tremendous deleterious mental health and socioeconomic impact of PTSD, research to understand and treat all aspects of PTSD is vitally important. One less recognized but highly significant consequence of PTSD is an increased risk of hypertension, cardiovascular disease (CV) disease, and its risk factors. Despite the epidemiologic data demonstrating increased CV risk in PTSD, very little is known about underlying mechanisms. This project will help fill this gap by examining the mechanistic role of sympathetic overactivation in PTSD. Sympathetic hyperactivity has a major role in causing and sustaining hypertension, and contributes to the development of heart failure, arrhythmias, and atherogenesis. Moreover, exaggerated SNS responses during mental stress are associated with an increased risk of hypertension and CV disease.

Slow breathing is an integral part of many ancient meditative practices that are purported to have beneficial physiologic and psychological effects. Clinical applicability of slow breathing requires a method for delivering slow breathing exercises to outpatients on a consistent basis. This can be achieved through device-guided slow breathing (DGB) in which breathing rate is slowed to < 10 breaths/min via an interactive biofeedback device. The RESPeRATE (Intercure, Inc.) device is currently FDA approved for adjunctive treatment of high blood pressure and reduction of stress. This device includes a belt-type respiratory sensor, earbuds to provide audio feedback, and microprocessor that measures adherence and success at achieving slow breathing rates.

Vagal nerve stimulation has been shown in both animal and human studies to safely and effectively reduce sympathetic activity and inflammation. tVNS is a noninvasive method that involves placing a device over the skin overlying the vagus nerve on the neck. The device delivers mild electrical stimulation, using transcutaneous electrical nerve stimulation (TENS) unit. Prior studies have shown that transcutaneous vagal nerve stimulation safely and effectively reduced muscle sympathetic nerve activity in healthy humans and improved heart rate variability, indicating a decrease in sympathetic nervous system (SNS) activity, and a shift in cardiac autonomic function toward parasympathetic (PNS) predominance.

The purpose of this study is to determine if device-guided slow breathing or tVNS improves sympathetic activity and vascular function in persons with PTSD. Participants will be randomized to 15 minutes daily of DGB vs sham-DGB, or tVNS vs. sham-tVNS for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* prehypertensive and normotensive veterans with PTSD, and prehypertensive and normotensive veterans without PTSD (controls)

Exclusion Criteria:

* heart or vascular disease
* illicit drug use within the last 6 months
* excessive alcohol use (>2 drinks per day)
* pregnancy
* autonomic dysfunction
* medications known to affect SNS (clonidine)
* treatment with monoamine oxidase (MAO) inhibitors within the last 14 days
* any serious systemic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-07 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in Muscle Sympathetic Nerve Activity (MSNA) Burst Frequency at Rest | Baseline, Week 8
  MSNA is assessed with microneurography where a tungsten microelectrode inserted in the nerve records sympathetic nerve activity.
Change in Baroreflex Sensitivity (BRS) at Rest | Baseline, Week 8
  Arterial baroreflex sensitivity (BRS) will be tested using pharmacologic manipulation of blood pressure at rest. BRS is assessed by measuring changes in MSNA and heart rate during arterial blood pressure changes induced by nitroprusside and phenylephrine.
Change in MSNA Burst Frequency While Under Mental Stress | Baseline, Week 8
  Mental stress will be induced by having participants complete mental arithmetic and with a combat virtual reality clip.
Change in BRS While Under Mental Stress | Baseline, Week 8
  Mental stress will be induced by having participants complete mental arithmetic and with a combat virtual reality clip. Arterial baroreflex sensitivity (BRS) will be tested using pharmacologic manipulation of blood pressure at rest and during mental stress.

SECONDARY OUTCOMES:
Endothelial Function | Baseline, Week 8
  Endothelial Function will be measured using peripheral arterial tonometry.
Vascular Stiffness | Baseline, Week 8
  Vascular stiffness will be measured noninvasively using pulse wave analysis and pulse wave velocity.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanie Park, MD, Principal Investigator — Emory University and the Atlanta VA Medical Center
Locations (1):
- Atlanta VA Medical Center, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fonkoue IT, Hu Y, Jones T, Vemulapalli M, Sprick JD, Rothbaum B, Park J. Eight weeks of device-guided slow breathing decreases sympathetic nervous reactivity to stress in posttraumatic stress disorder. Am J Physiol Regul Integr Comp Physiol. 2020 Oct 1;319(4):R466-R475. doi: 10.1152/ajpregu.00079.2020. Epub 2020 Aug 26. PMID 32847397